CLINICAL TRIAL: NCT04930835
Title: Treatment Outcomes With Full Arch Rehabilitations Supported by Immediate or Conventionally Loaded Implants: A Randomized Clinical Trial
Brief Title: Treatment Outcomes With Full Arch Rehabilitations Retained by Immediate or Conventionally Loaded Implants
Acronym: ILOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Full professor in Prosthodontics at the University of Salamanca, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ILOD
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Edentulous Jaw; Missing Teeth
MeSH Terms: conditions — Jaw, Edentulous; Anodontia | interventions — Dental Prosthesis, Implant-Supported

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Loading (Active Comparator): implants are loaded at least after two months of healing
  Interventions: Procedure: Implant supported dentures
- Immediate Loading (Experimental): implants are loaded the same day of surgery
  Interventions: Procedure: Implant supported dentures

INTERVENTIONS:
Procedure: Implant supported dentures — Placement of dental implants with different loading protocols for supporting full arch dentures.

SUMMARY:
This study aims to assess the treatment outcomes (clinical, functional and subjective) of full arch rehabilitations supported by implants with or without an immediate loading protocol. In this randomized clinical trial 20 fully edentulous patients were treated with full arch rehabilitations on dental implants. In half of the sample, the implants were loaded immediately by means of abutments after emplacement of the implant; but in the counterparts these abutments were connected to implants two months after the surgery (conventional protocol), and until that time the dentures were retained by healing abutments. Treatment outcomes were assessed at 2, 6 and 12 months after surgery. Clinical outcomes were quantified on the basis of implant failure rate, marginal bone loss and the peri-implant gingival index. Functional outcomes were calculated according to masticatory performance, estimated by the mixed fraction of a two-coloured chewing gum after 5, 10 and 15 chewing strokes, by the occlusal force recorded by pressure-sensitive sheets and by the bioelectrical muscular activity. The subjective outcomes of the treatment were assessed using both the oral satisfaction scale (visual analogue scale) and the Spanish version of the Oral Health Impact Profile (OHIP-20).

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous individuals who had lacked teeth for more than 10 years, routine users of conventional complete prostheses.
* sufficient amount of remaining bone to receive the implants in the region of the mandibular canines (minimum height=15 mm/minimum ridge width= 5mm)
* no evidence of systemic or psychic pathology that might contraindicate the implant treatment.

Exclusion Criteria:

* Those in which oral surgery or cognitive evaluations are contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Clinical Performance of Dental implants | One year after treatment
  Implant failure rate
Oral health-related quality of life | One year after treatment
  impact according to the OHIP-20 (Oral Health Impact Profile) instrument. The score range from 0 to 20, being 20 the worst outcome.
Mastication | One year after treatment
  Mixing ability tests
Area of Occlusal Occlusion | One year after treatment
  According to pressure-sensitive colorimetric sheets it is recorded the area in square millimeters
Occlusal Load | One year after treatment
  According to the pressure-sensitive colorimetric sheets , the load in both the anterior and posterior region of the arch are calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontológica de la Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No